CLINICAL TRIAL: NCT05527002
Title: Thoracic Endometriosis: A Cohort Study
Acronym: TORENDO
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Clinical Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 2509
Record Dates: First submitted 2022-05-01; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis Thoracic; Endometriosis of Lung; Endometriosis of Pleura; Endometriosis-related Pain; Endometriosis
Keywords: Medical therapy; Surgical treatment; Satisfaction
MeSH Terms: conditions — Endometriosis; Personal Satisfaction | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Satisfaction of patients after medical and surgical treatment for thoracic endometriosis — It is a retrospectively evaluation of cases of thoracic endometriosis in our clinic over the last 20 years, based on the review of medical records and on outpatient follow-up visits.
  The questionnaire are filled in routinely by patients attending the endometriosis center of this institute every 6 months. We will collect data relating to these questionnaires referring prospectively to the study period.
  If the questionnaires have not already been filled in by the patient, she will be contacted to fill them in, after signing the informed consent of the study.

SUMMARY:
Endometriosis is defined as the presence of endometrial glands and stroma outside the uterine cavity. It is an estrogen-dependent chronic inflammatory disease. Estimates show that up to 10% of premenopausal women have endometriosis. The most frequent forms of endometriosis are superficial peritoneal implants, ovarian cysts and deep nodules or plaques. However, the pelvis is not the exclusive site of endometriotic lesions: endometriosis can also affect the diaphragm, the pleura and the lung. All these localizations are included in the spectrum of "thoracic endometriosis".

Thoracic endometriosis may present with cough, wheezing, catamenial pneumothorax, hemothorax, hemoptysis and pulmonary nodules. If the diaphragmatic pleura is also involved, catamenial periscapular or neck pain may be associated with irritation of the phrenic nerve. The symptoms of thoracic endometriosis generally have catamenial onset. Thoracic endometriosis rarely occurs isolated. It is considered a progression of pelvic endometriotic disease. Due to its varied presentation, diagnosis can be particularly difficult and often only identified due to clinical suspicion. The instrumental diagnosis of pneumothorax and catamenial hemothorax can be obtained by radiography or computerized axial tomography of the chest. Magnetic resonance imaging is to be preferred in case of diaphragmatic involvement. The gold standard remains exploratory laparoscopy, possibly accompanied by Video Assisted Thoracic Surgery (VATS).

The first-line treatment is hormone therapy, aimed at suppressing ovulation and also preventing the onset of relapses. GnRH analogues are very effective in reducing the painful symptoms associated with endometriosis, but are not superior to other first-line treatments available. Furthermore, the prolonged hypoestrogenism can cause menopausal symptoms and osteoporosis.

Surgery should be considered a second-line treatment in case of intolerance or ineffectiveness of medical therapy. The surgical approach is multidisciplinary and involves the endoscopist gynecologist and the thoracic surgeon expert in VATS.

The principal aim of the study is the retrospective evaluation of thoracic endometriosis cases in our clinic over the last 20 years in order to evaluate the effectiveness of medical and surgical treatments in terms of satisfaction of patients suffering from this clinical condition. The secondary aim is to investigate the pathogenetic aspects of this clinical condition.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial glands and stroma outside the uterine cavity. It is an estrogen-dependent chronic inflammatory disease, in which the ectopic endometrium grows and proliferate under the action of estradiol. Estimates show that up to 10% of premenopausal women and 35% to 50% of women with infertility, pelvic pain or both, have endometriosis.

The most frequent forms of endometriosis are superficial peritoneal implants, ovarian cysts (endometrioma) and deep nodules or plaques (which can individually involve and infiltrate the parametria, Douglas pouch, anterior rectal wall, posterior vaginal fornix, antero-uterine pouch, bladder detrusor, ureters and sigmoid colon).

However, the pelvis is not the exclusive site of endometriotic lesions: endometriosis can also be localized outside the pelvis, resulting in the implantation and growth of an ectopic endometrium and catamenial symptoms.

In the thoracic cavity endometriosis can affect the diaphragm, the pleura and, ultimately, the lung. All these localizations are included in the spectrum of "thoracic endometriosis".

Thoracic endometriosis may present with cough, wheezing, catamenial pneumothorax, hemothorax, hemoptysis and pulmonary nodules. If the diaphragmatic pleura is also involved, catamenial periscapular or neck pain may be associated with irritation of the phrenic nerve.

Thoracic endometriosis rarely occurs isolated. It is considered a progression of pelvic endometriotic disease, due to the coexistence of pelvic localizations in up to 80% of cases and its onset at a later age (up to ten years later than pelvic endometriosis).

The diagnosis of thoracic endometriosis can be misleading, because the related symptoms can be very variable, from total asymptomaticity to catamenial pneumothorax (80%), catamenial hemothorax (14%), catamenial hemoptysis (5%) or, more rarely , appearance of pulmonary nodules.

The symptoms of thoracic endometriosis generally have catamenial onset (from 24 to 72 hours from the onset of menstrual flow), but can also appear remotely, in the event that the disease becomes chronic and the symptoms are linked to progressive clinical deterioration. Thoracic endometriosis involves the right hemithorax in 92% of cases and the left in 5% of cases; bilateral involvement occurs in only 3% of cases. Due to its varied presentation, diagnosis can be particularly difficult and often only identified due to clinical suspicion. The instrumental diagnosis of pneumothorax and catamenial hemothorax, exactly as for the non-catamenial equivalent, can be obtained by radiography or computerized axial tomography of the chest. Magnetic resonance imaging is to be preferred in case of diaphragmatic involvement; on the other hand, bronchoscopy is often not diagnostic because the endometriotic foci are located far from the mucous membranes of the main bronchi. The gold standard for the diagnosis of thoracic endometriosis remains exploratory laparoscopy, possibly accompanied by Video Assisted Thoracic Surgery (VATS). The evaluation of the presence of any diaphragmatic endometriotic implants should be routine during exploratory versus operative laparoscopy.

The first-line treatment is hormone therapy, aimed at suppressing ovulation. Medical therapy can also prevent the onset of relapses.

GnRH analogues are very effective in reducing the painful symptoms associated with endometriosis, but are not superior to other first-line treatments available. Furthermore, the prolonged hypoestrogenism can cause menopausal symptoms and osteoporosis.

Surgery should be considered a second-line treatment in case of intolerance or ineffectiveness of medical therapy. The surgical approach is multidisciplinary and involves the endoscopist gynecologist and the thoracic surgeon expert in minimally invasive surgery (VATS). Alternatively or to complete the excisional surgical treatment, in the case of pleural involvement, mechanical or chemical pleurodesis can be performed, which can reduce the risk of recurrence of pneumothorax by 20-25%.

The principal aim of the study is the retrospective evaluation of thoracic endometriosis cases in our clinic over the last 20 years in order to evaluate the effectiveness of medical and surgical treatments in terms of satisfaction of patients suffering from this clinical condition. Moreover, the secondary aim is to investigate the pathogenetic aspects of this clinical condition.

This is a case report, retrospective/prospective and monocentric study; it is based on the review of medical records and on outpatient follow-up visits of patients in our clinic with thoracic endometriosis. This is a study design that it is best suited to a low prevalence of disease.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50 years
* women with a diagnosis of thoracic endometriosis, in the presence or absence of other endometriotic localizations
* women referred to our tertiary-care endometriosis center " Fondazione IRCCS Ospedale Maggiore Policlinico", Milan, from 1 January 2000 to 01 March 2022.

Exclusion Criteria:

* the presence of concomitant diseases of the respiratory system
* women who denied their consensus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients referred to our endometriosis clinic and/or underwent surgery from 1 January 2000 to 01 March 2022 with a diagnosis of thoracic endometriosis were selected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied | 10 years
  a five-level Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied) to evaluate the effectiveness of medical and surgical treatments for thoracic endometriosis.
Number of patients greatly improved, much improved, minimally improved, unchanged, minimally worsened, very worsened and greatly worsened | 10 years
  Patients' Global Impression of Change (PGIC) scale, a composed of seven levels (greatly improved, much improved, minimally improved, unchanged, minimally worsened, very worsened, greatly worsened) to evaluate the effectiveness of medical and surgical treatments for thoracic endometriosis.
Number of patients with none, mild, moderate, severe or very severe symptoms | 10 years
  Patients' Global Impression of Severity (PGIS) scale, a scale consisting of five levels (none, mild, moderate, severe, very severe)
Mean scores of HADS- Hospital Anxiety and Depression Scale | 10 years
  The HADS questionnaire is a self-assessment mood scale specifically designed for use in non-psychiatric hospital outpatients to determine states of anxiety and depression. It comprises 14 questions, 7 for the anxiety subscale and 7 for the depression subscale.
  Lower scores indicate better psychological status
Mean scores of the Short Form Survey, SF-12 | 10 years
  The SF-12 health survey, developed from the original SF-36 questionnaire, is a well-known, validated, self-administered 12-item instrument. It measures health dimensions covering functional status, well-being, and overall health. Information from the 12 items is used to construct Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) measures, with higher scores indicating better health perception.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Berlanda, Prof, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy